CLINICAL TRIAL: NCT01701622
Title: The Blood Pressure Effects of Febuxostat in Patients Previously Treated With Allopurinol: A Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to enroll participants
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Deborah Minor, Pharm D, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0186
Record Dates: First submitted 2010-01-27; First posted 2012-10-05 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2017-12

CONDITIONS: Blood Pressure; Gout
Keywords: Blood Pressure; Gout; allopurinol; febuxostat; uric acid
MeSH Terms: conditions — Gout | interventions — Febuxostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allopurinol, febuxostat (Experimental): Patients currently treated with allopurinol will be switched to febuxostat, and the blood pressure differences between the two arms will be compared.
  Interventions: Drug: febuxostat

INTERVENTIONS:
Drug: febuxostat — If baseline allopurinol dose < 300 mg daily, will initiate febuxostat 40 mg daily.
  If baseline allopurinol dose > 300 mg daily, will initiate febuxostat 80 mg daily.
  Febuxostat is to be continued for 4 weeks, with blood pressure assessments by clinic and ambulatory blood pressure measurement at baseline and after 4 weeks.
  Other Names: Uloric

SUMMARY:
Hyperuricemia (high uric acid level) has been correlated to hypertension (high blood pressure) and overall cardiovascular disease risk in several studies. The relationship has even been noted to be independent of metabolic syndrome and kidney function. It has been repeatedly noted that hyperuricemia was an independent risk factor of death in those at high cardiovascular disease risk. A recent review concluded that there is strong evidence that hyperuricemia and gout are coupled with atherosclerosis and cardiovascular events.

Although this correlation of hypertension and hyperuricemia is known, there has only been one published study that has evaluated if lowering the uric acid would reduce the blood pressure. The authors concluded that in newly diagnosed hypertensive adolescents, allopurinol decreased the blood pressure. Despite this, further evaluation of this therapeutic approach has not been studied.

The hypothesis of this study is that febuxostat, a new xanthine oxidase inhibitor, has blood pressure lowering effects superior to allopurinol in patients diagnosed with gout.

DETAILED DESCRIPTION:
Screening and Recruitment

* Identify and recruit 20 participants from the University of Mississippi Medical Center General Internal Medicine/Hypertension and Family Medicine Clinics.
* Participants must be currently taking allopurinol for the treatment of gout and be on a stable dose of allopurinol for at least 2 months.
* Any antihypertensive medications must be at stable doses for at least 2 months.
* The identified patients will be invited to participate in the study.

Provide Consent

* IRB approved comprehension survey will be administered to participants in determination of competency to provide consent.
* The "Consent to Participate in Research" information will be discussed with each participant and consent acquired.
* Materials can be taken by the potential participant to review and consent provided at a later date.

Data collection

* After consent is provided, study personnel will evaluate blood pressure (BP).
* Participants will undergo 24-hour Ambulatory Blood Pressure Monitor (ABPM). The normal fee for ABPM will be waived.
* Participants will then discontinue allopurinol and initiate febuxostat at a comparable dose. Febuxostat will be provided to all participants at no cost.

  * If receiving < 300 mg allopurinol daily, will provide febuxostat 40 mg daily.
  * If receiving > 300 mg allopurinol daily, will provide febuxostat 80 mg daily.
* After at least 4 weeks of febuxostat, the participant will repeat 24-hour ABPM. The normal fee for ABPM will be waived.
* After completion of the febuxostat portion of the study, participants will receive a compensation of $50 at the end of the study. Compensation will only be provided to those who complete the entire study.

Results

* Data collection will be added to participant's permanent medical records.
* Results for individual participants will be discussed with the participant as well as their primary care provider.
* The decision to remain on febuxostat or resume allopurinol will lie with the primary care provider.

ELIGIBILITY:
Inclusion Criteria:

* Patients currently treated at the University of Mississippi Medical Center General Internal Medicine/Hypertension or Family Medicine Clinics.
* Have a diagnosis of gout.
* Taking allopurinol at a stable dose for at least 2 months.

Exclusion Criteria:

* Less than 18 years old.
* Severe renal impairment defined as CrCl <30 mL/min.
* Previous diagnosis of severe hepatic impairment.
* Currently taking azathioprine, mercaptopurine, or theophylline.
* Pregnant, breastfeeding, or anticipating pregnancy or breastfeeding.
* Arm circumference greater than 50 cm.
* Change in antihypertensive medication within the previous 2 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amber S Holdiness, PharmD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center General Medicine/Hypertension and Family Medicine Clinics, Jackson, Mississippi, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment - January 2010 - October 2011 Medical clinic
Pre-assignment Details: No significant events or approaches to report.
Groups:
- Allopurinol, Febuxostat: Patients currently treated with allopurinol will be switched to febuxostat, and the blood pressure differences between the two arms will be compared.
  febuxostat : If baseline allopurinol dose < 300 mg daily, will initiate febuxostat 40 mg daily.
  If baseline allopurinol dose > 300 mg daily, will initiate febuxostat 80 mg daily.
  Febuxostat is to be continued for 4 weeks, with blood pressure assessments by clinic and ambulatory blood pressure measurement at baseline and after 4 weeks.
Period: Overall Study
Arm/Group | Allopurinol, Febuxostat
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Allopurinol, Febuxostat
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1
Blood pressure [Mean (Standard Deviation); unit: mm Hg]
  Diastolic Blood Pressure | 79
  Systolic Blood Pressure | 131

OUTCOME MEASURES:

1. Primary Outcome: BP Differences While on Allopurinol and Febuxostat by Clinic Blood Pressure Readings and 24-hour Ambulatory Blood Pressure Readings
Description: The data collected will be analyzed and categorized according to age, race, gender, weight, height, 24-hour ABPM (24-hour systolic blood pressure (SBP)/diastolic blood pressure (DBP), trough SBP/DBP, and the mean nighttime SBP/SBP). Clinic systolic and diastolic BP and 24-hour AMBPs will be compared between the two treatments.
Time Frame: 4 to 5 weeks
Population: no analysis, as only one participant
Groups:
- Allopurinol, Febuxostat: Patients currently treated with allopurinol will be switched to febuxostat, and the blood pressure differences between the two arms will be compared.
  febuxostat: If baseline allopurinol dose < 300 mg daily, will initiate febuxostat 40 mg daily.
  If baseline allopurinol dose > 300 mg daily, will initiate febuxostat 80 mg daily.
  Febuxostat is to be continued for 4 weeks, with blood pressure assessments by clinic and ambulatory blood pressure measurement at baseline and after 4 weeks.
Arm/Group | Allopurinol, Febuxostat
Number analyzed (Participants) | 0

2. Secondary Outcome: If Patients With Hypertension Receive a Greater Reduction in Blood Pressure (BP) While on Febuxostat (Versus Allopurinol)
Description: measured by mean 24-hour systolic blood pressure (SBP)/diastolic blood pressure (DBP), trough SBP/DBP, and mean nighttime SBP/SBP while on allopurionol and febuxostat.
Time Frame: Participants will be followed for an expected average of 4 to 5 weeks.
Groups:
- Allopurinol, Febuxostat: Patients currently treated with allopurinol will be switched to febuxostat, and the blood pressure differences between the two arms will be compared.
  febuxostat: If baseline allopurinol dose < 300 mg daily, will initiate febuxostat 40 mg daily.
  If baseline allopurinol dose > 300 mg daily, will initiate febuxostat 80 mg daily.
  Febuxostat is to be continued for 4 weeks, with blood pressure assessments by clinic and ambulatory blood pressure measurement at baseline and after 4 weeks.
  as reported earlier (2013), no statistical analysis because of no study participate completion
Arm/Group | Allopurinol, Febuxostat
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: adverse event data collected over a total period of 4 weeks
Description: Spontaneously report adverse events
Groups:
- Febuxostat: Febuxostat group. The primary outcome of the study is the 24 hour ABPM differences while participants were taking allopurinol compared to taking febuxostat.
Arm/Group | Febuxostat
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Early termination leading to no subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes